CLINICAL TRIAL: NCT00738543
Title: Comparative Study of 10% Povidone-iodine Against 10% Sodium Hypochlorite as Skin Antiseptics in Human Volunteers.
Brief Title: Povidone-iodine Against Sodium Hypochlorite as Skin Antiseptics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad de Guanajuato (Other)
Collaborators: Concejo de Ciencia y Tecnología del Estado de Guanajuato (Unknown); Pisa SA de CV (Unknown)
Responsible Party: Principal Investigator, Alejandro E. Macias, Profesor de tiempo completo, Universidad de Guanajuato
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: FMUGAmuch
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Results first posted 2010-08-17 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2009-02

CONDITIONS: Healthy Volunteers
Keywords: Antiseptics; Administration, cutaneous; Iodophors; Chlorine compounds; Anti-infecting agents, local
MeSH Terms: interventions — Povidone-Iodine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Whole group of 48 volunteers (Experimental): The arm is composed of 48 human volunteers to test 10% povidone-iodine (Isodine Solucion ®, Boehringer-Ingelheim Promeco, Mexico City), Hypochlorite 10% of electrochemical production (Exsept 10% ®, Pisa, Guadalajara, Mexico), and control.
  Interventions: Other: WHOLE GROUP OF 48 VOLUNTEERS

INTERVENTIONS:
Other: WHOLE GROUP OF 48 VOLUNTEERS — Two antiseptics (10% povidone iodine and 10% sodium hypochlorite) and one control were tested as skin antiseptics. The intervention consisted of preparing the skin with the antiseptic or the control. The areas were approximately 25 cm2 on the forearm for each antiseptic or control. The antiseptic or control were applied in an outward circular motion using a swab that was soaked with the solution. The solution was then kept on the skin for 60 seconds before the bacterial culture was conducted. All volunteers were instructed to continue the use of neutral soap and shampoo without antiseptics during the follow-up period.
  Other Names: Isodine (R); Exsept (R)

SUMMARY:
The investigators have few options for skin antisepsis. Alternatives for povidone-iodine, which is the most commonly used agent, are costly or ineffective. To have more options, this study is needed. The investigators want to know if there are difference between the use of 10% sodium hypochlorite or 10% povidone-iodine for skin antisepsis.

DETAILED DESCRIPTION:
Sodium hypochlorite at 10% has been widely used as antiseptic in patients on dialysis as well as for irrigation of wounds and burns. Since it has been used successfully in caring for the exit site of hemodialysis catheters, it is reasonable to propose its use for the insertion and care of central intravascular catheters, as well as for skin preparation before surgery. Alternatives for povidone-iodine, which is the agent most commonly used, are costly or ineffective. To have more options, this study is needed to know if 10% sodium hypochlorite is similar to the most common option for skin antisepsis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers.

Exclusion Criteria:

* History of skin allergies or atopy, as well as reactions to soaps, iodine, chlorine, or latex

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro E Macias, M. D., Principal Investigator — Universidad de Guanajuato
Locations (1):
- University of Guanajuato School of Medicine, León, Guanajuato, Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers recruited from August to December 2008 in the Microbiology Laboratory of University of Guanajuato, Mexico.
Pre-assignment Details: For stabilization of skin microbiota, all volunteers used neutral soap and shampoo without antiseptics over a period of two weeks, being advised to avoid swimming in pools.
Groups:
- Whole Group: Human volunteers to test control, povidone-iodine and hypochlorite as skin antiseptics
Period: Povidone Iodine
Arm/Group | Whole Group
Started | 48
Completed | 48
Not Completed | 0
Period: Sodium Hypochlorite
Arm/Group | Whole Group
Started | 48
Completed | 48
Not Completed | 0
Period: Control
Arm/Group | Whole Group
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Whole Group
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 24.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 24
Region of Enrollment [Number; unit: participants]
  Mexico | 48

OUTCOME MEASURES:

1. Primary Outcome: Bacterial Count of Skin Cultures for the 10% Povidone-iodine Period
Description: Bacterial colony count of skin cultures to determine antiseptic properties
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: Colony-forming units per cm squared
Arm/Group | Whole Group
Number analyzed (Participants) | 48
Colony-forming units per cm squared | 231 [77 to 615]
Statistical Analysis 1: Comparison: Whole Group; The null hypothesis established that the three medians were equal. To test significant differences for non-normally distributed data, a range test (Kruskal-Wallis) was used; Test type: Non-Inferiority or Equivalence — A minimal sample of 20 volunteers was calculated to to find a difference of 200 CFU/mL, with a power of 80% and bilateral error of 5%; p < 0.05, Kruskal-Wallis — Post-hoc test of Kruskal-Wallis for multiple comparisons of Z values was used to determine which arm was different; 2 degrees of freedom corrected for ties

2. Secondary Outcome: Presence of Skin Reactions for the 10% Povidone-iodine Period
Description: Presence of allergy or any skin reaction at 24 hours after the antiseptic application
Time Frame: 24 hours
Population: A minimal sample of 20 volunteers was calculated to find a difference of 200 CFU/mL, with a power of 80%, and bilateral error of 5%. Analysis per protocol.
Measure: Number; unit: Number of participants with skin reactio
Arm/Group | Whole Group
Number analyzed (Participants) | 48
Number of participants with skin reactio | 0

3. Primary Outcome: Bacterial Colony Forming Units for the 10% Sodium Hypochlorite Period
Description: After incubation, the outcome assessor counted the colonies to determine the colony-forming units per square centimeter (CFU/cm2) of skin.
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: Colony-forming units per cm squared
Arm/Group | Whole Group
Number analyzed (Participants) | 48
Colony-forming units per cm squared | 192 [77 to 519]
Statistical Analysis 1: Comparison: Whole Group; The null hypothesis established that the 3 medians were equal. To test significant differences for non-normally distributed data, a range test (Kruskal-Wallis) was used. The alpha level for significance was established at 5%. A minimal sample of 20 volunteers was calculated for a power of 80%, and bilateral error of 5%; Test type: Non-Inferiority or Equivalence — The minimal sample of 20 volunteers was calculated to find a difference of 200 CFU/mL; p < 0.05, Kruskal-Wallis — Post-hoc test of Kruskal-Wallis for multiple comparisons of Z values was used to determine which arm was different; 2 degrees of freedom corrected for ties

4. Primary Outcome: Bacterial Colony Forming Units for the Control Period
Description: as for outcome 3
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: Colony-forming units per cm squared
Arm/Group | Whole Group
Number analyzed (Participants) | 48
Colony-forming units per cm squared | 1500 [635 to 3269]

5. Secondary Outcome: Presence af Allergy or Skin Reaction for the 10% Sodium Hypochlorite Period
Description: Presence of allergy or skin reaction at 24 hours after the application of the antiseptic
Time Frame: 24 hours
Measure: Number; unit: Number of participants with reaction
Arm/Group | Whole Group
Number analyzed (Participants) | 48
Number of participants with reaction | 0

ADVERSE EVENTS:
Time Frame: 24 hours following the application of the antiseptics or control
Description: All the participants were at risk for non-serious adverse events, "0" means that none suffered any adverse event.
Arm/Group | Whole Group
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No